CLINICAL TRIAL: NCT01095354
Title: Investigation of Lung Ventilation Inhomogeneity in Pediatric Asthma: Multiple Breath Washout and Asthma
Brief Title: Investigation of Lung Ventilation Inhomogeneity in Pediatric Asthma
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Padmaja Subbarao, Staff Respirologist, The Hospital for Sick Children
Other Study IDs: 1000013927
Record Dates: First submitted 2010-03-23; First posted 2010-03-30 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: pediatric; lung ventilation inhomogeneity
MeSH Terms: conditions — Asthma | interventions — Salts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples will be processed and divided into two categories: eosinophilic (% eosinophils >2.5%) and non-eosinophilic (<2.5% eosinophils). The two categories of asthmatics will be used to categorize asthmatics for comparison on parameters such as SnIII analysis of SF6, LCI etc. In addition, % eosinophilia will be considered as a continuous measure in those with % eosinophils > 2% and correlated with LCI.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma Patients: Spirometry. Bronchodilator with Salbutamol. Induced sputum in > 10 years of age using Sodium Chloride Inhalation. Multiple Breath Washout (MBW).
  Interventions: Drug: Sodium Chloride Inhalation

INTERVENTIONS:
Drug: Sodium Chloride Inhalation — Spirometry: all subjects Plethysmography and exhaled nitric oxide: >6 years Multiple Breath Washout: Tidal breathing using a facemask <9 years or mouthpiece >9 years. Wash-in phase: gas mixture containing 4% SF6, 4% He, 21% oxygen and balance nitrogen inhaled until steady state. Bias flow stopped during expiration by removal of T-piece. Wash-out phase: patient inspires room air and exhales tracer gas until SF6 reaches <0.1%.
  Bronchodilator response: Bronchodilator (Salbutamol 400 mcg) to asthma subjects, spirometry and MBW repeated after 15 minutes.
  Induced sputum in asthma subjects >10 yrs. Post-bronchodilator spirometry, subject inhales concentrations of 3, 4 and 5% hypertonic saline for 7 minutes for 3 cycles until expectorating sputum.
  Other Names: Salt, NaCl

SUMMARY:
The primary objective of this study is to determine if well-controlled asthmatic patients followed in subspecialty asthma clinics between the ages of 3 - 18 years can be distinguished from healthy controls using lung clearance index, a parameter from the multiple breath washout test. Also, to correlate lung clearance index with asthma sputum cell counts.

DETAILED DESCRIPTION:
Clinical studies are underway which are examining the utility of the LCI in obstructive respiratory disease (cystic fibrosis and asthma). However, the majority of studies have examined asthmatics with ongoing evidence of reversible disease on spirometry. There is a very limited body of research comparing LCI values in well-controlled asthmatics to healthy controls. Furthermore, the type of inflammation occurring in asthma may have a different site of action, we will prospectively study whether there is a difference in LCI between eosinophilic and neutrophilic inflammation to give us an indication of whether the site of non-eosinophilic inflammation is primarily in the small airways as well.

ELIGIBILITY:
Inclusion Criteria:

* Asthma Subjects:

  * 3 - 18 years of age at enrolment
  * Clinically stable at enrolment
  * Physician diagnosis of asthma and attending follow-up in the Asthma Clinic

Exclusion Criteria:

* Asthma Subjects:

  * Born premature (before 37 weeks gestational age)
  * Low birth weight (less than 2.5 kilograms)
  * History of congenital heart disease, neuromuscular disorder or bone disease
  * History of any chronic lung disease other than asthma
  * Respiratory infection in last three weeks
  * Change in medication in last three weeks (including oral steroids)
  * Current or previous history of smoking

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Asthma patients will be recruited from the Respiratory Medicine clinic at the Hospital for Sick Children. A member of the medical team in the Asthma Clinic, known to the patient, will introduce the study, and obtain permission for the patient/caregiver to meet with study personnel. Subjects will then be approached by the Principal investigator or her delegate. They will be informed that enrolment is voluntary and that they can withdraw from the study at any time.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Lung Clearance Index (LCI) | Day 1
  Lung clearance index will be compared between healthy and asthmatic patients after they have performed Pulmonary Function Testing and Multiple Breath Washout

SECONDARY OUTCOMES:
Correlation of sputum cell counts with LCI | Day 1
  Sputum induction for specimen collection
Effect of bronchodilator on baseline and post-spirometry LCI | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Padmaja Subbarao, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
scientific journal articles